CLINICAL TRIAL: NCT01668979
Title: Assessment of a New System to Detect, Quantify and Treat Near Falls in Older Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Director of Research and Development, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-12-NG-0363-CTIL
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Idiopathic Fallers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- new system to detect Near Falls: the new system comprises of a treadmill and a virtual reality simulation that will be used to induce Near Falls in healthy older adults with a history of falls.
  Interventions: Device: new system to detect Near Falls

INTERVENTIONS:
Device: new system to detect Near Falls — We will invite healthy older adults with a history of falls to try the new system and assess whether the new system can induce, detect and quantify Near Fall episodes

SUMMARY:
The study is aimed to assess a new system for the automatic detection, quantification and treatment of Near Fall (NF) episodes in healthy older adults with a history of falls. The system is comprized of a treadmill and a virtual reality simulation which provides a motor-cognitive challenge to provoke NF. The challenges provided by the system are individualized and using machine learning algorithms will enable the identification and detection of NF under different conditions and allow for the most suitable treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy older adults with a history of falls or complaints of gait instability
2. Able to walk independently for at least 10 minutes

Exclusion Criteria:

1. Systemic chronic or acute pathologies:

   1. Ischemic heart disease
   2. Orthopedic or Rheumatic diseases
   3. Severe vision problems
   4. Neurological disease: PD, AD, CVA
2. Patients who underwent brain surgery in the last 6 months prior to the study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older adults with a history of falls
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
usability of the system to detect Near Falls | one year

SECONDARY OUTCOMES:
Near Fall severity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel